CLINICAL TRIAL: NCT03569488
Title: Validation of the French Version of the Low Anterior Resection Syndrome (LARS) Score for Measuring Bowel Dysfunction After Sphincter-preserving Surgery Among Rectal Cancer Patients
Brief Title: Validation of the French Version of the Low Anterior Resection Syndrome (LARS) Among Rectal Cancer Patients
Acronym: LARS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: National Cancer Institute, France (Other Government); French Research Group of Rectal Cancer Surgery (GRECCAR) (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 17-247
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Rectal Cancer Patients
Keywords: quality of life; sphincter-sparing surgery; LARS score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FT-LARS questionnaire — FT-LARS questionnaire

SUMMARY:
Oncological rectal cancer outcomes have improved considerably because of optimal surgery by total mesorectal excision in conjunction with multidisciplinary team management by selective multimodal therapy (ie, neo-adjuvant chemo-radiotherapy). The 5-year survival has increased to more than 50% and local recurrence has been reduced to less than 10%. These advancements have resulted in more patient receiving sphincter-preserving surgery (SPS). With an increasing number of rectal cancer survivors, the investigators observe a rising attention to the disordered bowel function after SPS, called "low anterior resection syndrome" (LARS). LARS appear immediately after surgery, becoming most pronounced during the first few months, and improved thereafter, reaching a steady state after around two years. However, up to 60% of patients with SPS suffer from LARS which impaired their quality of life (QoL). The prevalence and severity of LARS is difficult to assess due to heterogeneity of the assessment tools. A group of Danish authors have recently developed and validated a five-item instruments for evaluation of LARS (LARS score). It represents to date the best questionnaire to capture anorectal postoperative function and consists of five items: incontinence for flatus, incontinence for liquid stool, frequency of bowel movements, clustering of stools, and urgency. It allows a categorization of patients into 3 groups: no LARS (0-20 points), minor LARS (21-29 points), and major LARS (30-42 points). Developed in Danish, it is now internationally validated with translations in Chinese, English, German, Spanish and Swedish. To our knowledge, French version of the LARS score is not yet available. The aim of our study will be to adapt the LARS scale questionnaire to the French language (LARS-F), and assess its psychometric properties.

Inclusion criteria will be patients 18 years old or above who were operated for rectal cancer from 2007 to 2015. Exclusion criteria will include the presence of stoma and/or known disseminated or recurrent disease. Patients will be identified through local databases by the local investigators at each of the participating centers with a minimum duration of 24 months after surgery to allow their bowel function to have regained stability. This study will be supported by the French Research Group of Rectal Cancer Surgery in order to allow the feasibility of the project.

After translation/back-translation procedures in accordance with the permission from the original authors, the LARS-F score and the whole translation process will be then sent to the original authors for approval. Then a pilot study will be conducted. The French questionnaire (LARS-F score) will be then administered to 100 patients in order to verify the adequacy and degree of comprehension of the questions. Reproducibility will be investigated by a test-retest procedure. A randomly selected subgroup of participants (n= 400) will be sent the LARS-F score questionnaire twice (with an interval of two weeks). The test-retest reliability of the questionnaire will be assessed by the Cohen's Kappa (no, minor and major LARS scores) or by intra-class correlation coefficient, ICC (quantitative LARS score). Then, eligible patients will receive a postal invitation to complete the LARS-F score and the l'European Organization for Research and treatment of Cancer (EORTC) QLQ-C30 and QLQ-CR29, respectively. The validity of the LARS-F score will be tested by using the indicators of convergent validity and discriminant validity. The convergent validity will be determined notably in this study by computing the correlations between the LARS-F score and the EORTC QLQ-C30 and QLQ-CR29 domains. For discriminant validity testing, the investigators will use known variables to affect bowel function after SPS, such as gender, age, neo-adjuvant radiation therapy, distance of the tumor from the anal verge, prior temporary stoma, and length of postoperative period.

The validation of the French version of the LARS score will allow to use a scientific instrument in order to assess both prevalence and severity of LARS. This instrument will allow to develop a future research and clinical practice in France. It will be used in the daily clinical practice to identify patients with LARS score. It will hopefully lead to improve the awareness of clinicians, in order to improve the prevention and the treatment of bowel dysfunction, as well as the information given to patients. In the future, the investigators will able to develop a new patient-led follow-up program based on symptom burden and health-related QoL.

DETAILED DESCRIPTION:
Inclusion Criteria:

* Age between 18 and 80 years
* Rectal cancer patients undergoing curative sphincter-preserving surgery with partial or total mesorectal excision
* Surgery performed between January 2007 to January 2016, with reversal of the defunctioning stoma before January 2016;
* Hence all patients had had bowel continuity restored for at least 24 months Voluntarily participated in the study

Exclusion Criteria:

* The presence of stoma and/or known disseminated or recurrent disease
* Other diseases of bowel dysfunction (Crohn's disease)
* Cognition and/or language issues.

Detailed description of the implemented techniques

-The validation study of the French version of the LARS score is based on one hand on the face and content validities and on the other hand on the measurement of its psychometric properties in compliance with the standards published by American Educational Research Association & al.

Outcomes measures

* After translation/back-translation procedures in accordance with the permission from the original authors, the LARS-F score and the whole translation process will be then sent to the original authors for approval. Then, eligible patients will receive a postal invitation to complete the LARS-F score and the l'European Organization for Research and treatment of Cancer (EORTC) QLQ-C30 and QLQ-CR29, respectively. For each item, ceiling and floor effects will be sought.
* The reliability will be assessed by both internal consistency (Cronbach's alpha coefficient).
* To evaluate reproducibility, a test-retest study will be performed in a randomly selected subgroup patients by comparing LARS-F scores obtained between the patient's first and second postal invitation (in an interval of 7-14 days).
* The correlations between the LARS-F score and the EORTC QLQ-C30 and QLQ-CR29 domains will allow to determine convergent validity. For discriminant and divergent validities testing, we will hypothesize that the LARS score will differentiate between the bowel functions of patients with different demographic or clinical features such as sex, age, length of postoperative period, distance of the tumor from the anal verge, radiation therapy, and prior temporary stoma.
* Sensitivity and specificity for minor and major LARS scores will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Rectal cancer patients undergoing curative sphincter-preserving surgery with partial or total mesorectal excision
* Surgery performed between January 2007 to January 2016, with reversal of the defunctioning stoma before January 2016;
* Hence all patients had had bowel continuity restored for at least 24 months Voluntarily participated in the study

Exclusion Criteria:

* The presence of stoma and/or known disseminated or recurrent disease
* Other diseases of bowel dysfunction (Crohn's disease)
* Cognition and/or language issues.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2020-01-24 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
validation of the French version of the LARS score | baseline
  * Cross cultural adaptation
  * Reliability :
    * Test-retest
    * Internal consistency
  * Face validity and content validity
  * Floor effect - Ceiling effect
  * Discriminant validity
    * Convergent validity and Divergent validity
    * Known-group method and relationship between each item and subscales

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Chru Amiens, Amiens
  - Caen University Hospital, Caen
  - Chru Lille, Lille
  - Centre Oscar Lambret, Lille
  - Chru Nancy, Nancy
  - Chru Nantes, Nantes
  - Chru Tours, Tours
  - clc VANDEUVRE LES NANCY, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Sarcher T, Dupont B, Alves A, Menahem B. Anterior resection syndrome: What should we tell practitioners and patients in 2018? J Visc Surg. 2018 Oct;155(5):383-391. doi: 10.1016/j.jviscsurg.2018.03.006. Epub 2018 Aug 17. PMID 30126800
- [Background] Abdelli A, Tillou X, Alves A, Menahem B. Genito-urinary sequelae after carcinological rectal resection: What to tell patients in 2017. J Visc Surg. 2017 Apr;154(2):93-104. doi: 10.1016/j.jviscsurg.2016.10.002. Epub 2017 Feb 1. PMID 28161008
- [Background] Rullier E, Rouanet P, Tuech JJ, Valverde A, Lelong B, Rivoire M, Faucheron JL, Jafari M, Portier G, Meunier B, Sileznieff I, Prudhomme M, Marchal F, Pocard M, Pezet D, Rullier A, Vendrely V, Denost Q, Asselineau J, Doussau A. Organ preservation for rectal cancer (GRECCAR 2): a prospective, randomised, open-label, multicentre, phase 3 trial. Lancet. 2017 Jul 29;390(10093):469-479. doi: 10.1016/S0140-6736(17)31056-5. Epub 2017 Jun 7. PMID 28601342
- [Background] Lakkis Z, Manceau G, Bridoux V, Brouquet A, Kirzin S, Maggiori L, de Chaisemartin C, Lefevre JH, Panis Y; French Research Group of Rectal Cancer Surgery (GRECCAR) and the French National Society of Coloproctology (SNFCP). Management of rectal cancer: the 2016 French guidelines. Colorectal Dis. 2017 Feb;19(2):115-122. doi: 10.1111/codi.13550. PMID 27801543
- [Background] Pieniowski EHA, Palmer GJ, Juul T, Lagergren P, Johar A, Emmertsen KJ, Nordenvall C, Abraham-Nordling M. Low Anterior Resection Syndrome and Quality of Life After Sphincter-Sparing Rectal Cancer Surgery: A Long-term Longitudinal Follow-up. Dis Colon Rectum. 2019 Jan;62(1):14-20. doi: 10.1097/DCR.0000000000001228. PMID 30394987
- [Background] Battersby NJ, Bouliotis G, Emmertsen KJ, Juul T, Glynne-Jones R, Branagan G, Christensen P, Laurberg S, Moran BJ; UK and Danish LARS Study Groups. Development and external validation of a nomogram and online tool to predict bowel dysfunction following restorative rectal cancer resection: the POLARS score. Gut. 2018 Apr;67(4):688-696. doi: 10.1136/gutjnl-2016-312695. Epub 2017 Jan 23. PMID 28115491
- [Background] Juul T, Ahlberg M, Biondo S, Espin E, Jimenez LM, Matzel KE, Palmer GJ, Sauermann A, Trenti L, Zhang W, Laurberg S, Christensen P. Low anterior resection syndrome and quality of life: an international multicenter study. Dis Colon Rectum. 2014 May;57(5):585-91. doi: 10.1097/DCR.0000000000000116. PMID 24819098
- [Background] Juul T, Ahlberg M, Biondo S, Emmertsen KJ, Espin E, Jimenez LM, Matzel KE, Palmer G, Sauermann A, Trenti L, Zhang W, Laurberg S, Christensen P. International validation of the low anterior resection syndrome score. Ann Surg. 2014 Apr;259(4):728-34. doi: 10.1097/SLA.0b013e31828fac0b. PMID 23598379
- [Background] Emmertsen KJ, Laurberg S. Low anterior resection syndrome score: development and validation of a symptom-based scoring system for bowel dysfunction after low anterior resection for rectal cancer. Ann Surg. 2012 May;255(5):922-8. doi: 10.1097/SLA.0b013e31824f1c21. PMID 22504191
- [Background] Juul T, Elfeki H, Christensen P, Laurberg S, Emmertsen KJ, Bager P. Normative Data for the Low Anterior Resection Syndrome Score (LARS Score). Ann Surg. 2019 Jun;269(6):1124-1128. doi: 10.1097/SLA.0000000000002750. PMID 31082911
- [Derived] Eid Y, Bouvier V, Dejardin O, Menahem B, Chaillot F, Chene Y, Dutheil JJ, Juul T, Morello R, Alves A. 'French LARS score': validation of the French version of the low anterior resection syndrome (LARS) score for measuring bowel dysfunction after sphincter-preserving surgery among rectal cancer patients: a study protocol. BMJ Open. 2020 Mar 8;10(3):e034251. doi: 10.1136/bmjopen-2019-034251. PMID 32152168